CLINICAL TRIAL: NCT03465111
Title: An Open Label, Multi-centered, Randomized Phase 2 Study to Evaluate the Safety, Tolerability and Bioactivity of Subcutaneous ACTH GeL in PAtients With Scleritis: The ATLAS Study
Brief Title: A Clinical Study to Evaluate the Potential Role of ACTH Gel in Patients With Scleritis
Acronym: ATLAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Metropolitan Eye Research & Surgery Institute (Other)
Collaborators: Mallinckrodt (Industry); Stanford University (Other); Ocular Imaging Research and Reading Center (Other); Foresight Studies, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #4301
Record Dates: First submitted 2018-02-16; First posted 2018-03-14 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Scleritis
Keywords: Scleritis; anterior; adrenocorticotropic hormone; ACTH; Non-infectious
MeSH Terms: conditions — Scleritis | interventions — Adrenocorticotropic Hormone; Gels

STUDY DESIGN:
Intervention Model Description: ATLAS is an Investigator-initiated, open-labelled, multi-center, randomized, phase II clinical trial, to evaluate the effect of two dose regimens of subcutaneous ACTH gel in subjects with non-infectious anterior scleritis. Thirty (30) subjects with non-infectious anterior scleritis will be enrolled and randomized (1:1) at their first visit to one of the two treatment arms:
  1. Mandatory 80 U twice weekly treatment with SC ACTH gel, starting at the Baseline visit (Day 0) until end of week 16. Starting at week 17, the treatment will be administered on as needed basis, based on the retreatment criteria.
  2. Mandatory 80 U thrice weekly treatment with SC ACTH gel, starting at the Baseline visit (Day 0) until end of week 16. Starting at week 17, the treatment will be administered on as needed basis, based on the retreatment criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Twice Weekly Treatment Arm (Experimental): Patients in this treatment arm will receive mandatory 80 U twice weekly treatment with SC ACTH (adrenocorticotropic hormone) gel, starting at the Baseline visit (Day 0) until end of week 16. Starting at week 17, the treatment will be administered on as needed basis, based on the retreatment criteria.
  Interventions: Drug: ACTH (adrenocorticotropic hormone) gel
- Thrice Weekly Treatment Arm (Experimental): Patients in this treatment arm will receive mandatory 80 U thrice weekly treatment with SC ACTH (adrenocorticotropic hormone) gel, starting at the Baseline visit (Day 0) until end of week 16. Starting at week 16, the treatment will be administered on as needed basis, based on the retreatment criteria.
  Interventions: Drug: ACTH (adrenocorticotropic hormone) gel

INTERVENTIONS:
Drug: ACTH (adrenocorticotropic hormone) gel — The dose of H.P. Acthar Gel is 80 Units administered subcutaneously
  Other Names: H.P. Acthar® Gel

SUMMARY:
ATLAS study is a clinical trial to evaluate the potential role of subcutaneous adrenocorticotropic hormone (ACTH) gel in the management of non-infectious scleritis.

Specifically, the ATLAS Study aims to evaluate the safety, tolerability and effect of 2 different dose regimens of ACTH gel administered by subcutaneous (SC) injection in patients with scleritis, over a period of 12 months.

Scleritis is an inflammatory disease affecting the sclera (white outer coating of the eye), which causes blurring of vision, redness, tearing and painful ocular inflammatory episodes in one or both eyes. Scleritis may results in vision threatening ocular complications, if left untreated. Treatment of scleritis is usually chronic and requires systemic therapy with non-steroidal anti-inflammatory drugs, corticosteroids and immunosuppressive therapy. Due to its treatment resistance nature, scleritis remains a therapeutic challenge for many ophthalmologists.

H.P. Acthar Gel (ACTH Gel) is a highly purified preparation of adrenocorticotropic hormone (ACTH) in a gel that is designed to provide extended release of the ACTH following injection. It is a FDA approved treatment for flares or on a regular basis (maintenance) in people with systemic lupus erythematosus (lupus), infantile spasms, adults with acute relapses or flares of multiple sclerosis (MS), patients with kidney diseases, among other indications. ACTH Gel is also approved for a wide range of allergic and inflammatory diseases of the eye.

Given the established role of inflammation in the pathogenesis of scleritis and the anti-inflammatory effects of ACTH Gel treatment by blocking various inflammatory pathways, a beneficial outcome could be anticipated from ACTH Gel treatment in patients with scleritis.

DETAILED DESCRIPTION:
ATLAS is an Investigator-initiated, open-labelled, multi-center, randomized, phase II clinical trial, to evaluate the effect of two dose regimens of subcutaneous ACTH gel in subjects with non-infectious anterior scleritis over a period of 12 months (52 weeks), with the primary endpoint at month 4 (week 16). ATLAS study will be conducted at up to 6 clinical sites in USA. The study will be coordinated by the Ocular Imaging Research and Reading Center (OIRRC), which will serve as the coordinating and reading center for the ATLAS Study.

The ATLAS Study aims to evaluate the potential role of subcutaneous adrenocorticotropic hormone (ACTH) gel, in the management of non-infectious anterior scleritis. Specifically, the ATLAS Study aims to evaluate the safety and tolerability of 2 different dose regimens of ACTH gel administered by subcutaneous (SC) injection in patients with non-infectious anterior scleritis and to evaluate the bioactivity of 2 different dose regimens of ACTH gel administered by SC injection in patients with non-infectious anterior scleritis.

Scleritis refers to red and painful inflammation, centered in the sclera that may involve adjacent ocular structures including the cornea, episclera and uvea. Scleritis may results in vision threatening ocular complications (corneal ulceration, cataract, glaucoma, retinal detachment, choroidal effusion) and subsequent blindness. Up to 50% of patients with scleritis have an associated systemic inflammatory disorder, such as sarcoidosis, rheumatoid arthritis, systemic lupus erythematosus, and polyangiitis with granulomatosis. Scleritis is classified based on the anatomic site, as anterior or posterior, with 90% of cases anterior. Anterior scleritis may manifest as necrotizing or non-necrotizing. Non-necrotizing, noninfectious scleritis is the most prevalent form. The course of scleritis is usually chronic, similar to uveitis, and requires systemic therapy with non-steroidal anti-inflammatory drugs and glucocorticoids, along with immunosuppression, as steroid-sparing therapy. Due to its treatment resistance nature, scleritis remains a therapeutic challenge for many ophthalmologists. The ultimate goal is to control the inflammation, which serves as the cornerstone of the scleritis pathophysiological basis.

Adrenocorticotropic hormone (ACTH) is a member of a group of peptide hormones, called melanocortins (MCs). ACTH is released from the pituitary gland and acts primarily on the adrenals to stimulate and regulate steroid hormones production. It has been demonstrated that MCs can be produced by immune cells at the inflammation site, which created a special interest in immunomodulatory properties of these peptides. Latest evidence proposes other anti-inflammatory mechanisms of ACTH actions in addition to steroidogenesis, including leukocyte transmigration inhibition, cytokine synthesis reduction and generation of anti-inflammatory signals locally at the inflammation site. ACTH gel has been reported to be effective in various systemic inflammatory diseases including nephrotic syndrome, multiple sclerosis, opsoclonus myoclonus,dermatomyositis and polymyositis. These reports also include cases that were resistant to steroids and other immunomodulatory drugs, supporting the immune-modulating properties of ACTH. H.P. Acthar® Gel (Repository Corticotropin Injection, Mallinckrodt Pharmaceuticals) is a 39-amino-acid, pituitary-derived ACTH analogue. ACTH gel has been demonstrated to have additional therapeutic effects on the humoral immune system, independent of its role in the adrenal steroidogenesis regulation. It is approved by the US FDA for treatment of a number of inflammatory conditions, including multiple sclerosis, rheumatic and collagen disorders, as well as ophthalmologic diseases, such as ocular allergy, keratitis, uveitis and optic neuritis. However, due to the scarcity of data from clinical studies, many physicians are unaware of ACTH gel as a treatment option for inflammatory diseases.

The proposed study aims to evaluate the potential role of ACTH gel in the management of non-infectious anterior scleritis. Given the established role of inflammation in the pathogenesis of scleritis and the ability of ACTH to bind to cellular and tissue melanocortin receptors, thus blocking various inflammatory pathways, a beneficial outcome could be anticipated from ACTH analogue in patients with scleritis.

Thirty (30) subjects with non-infectious anterior scleritis will be enrolled in the study.

The primary endpoint of the study will be at week 16, with an active, as-needed treatment extension phase from week 17 to week 52.

All study participants will be randomized (1:1) at their Baseline (BL) visit (visit 2) to one of the two treatment arms. All subjects will be started on oral corticosteroids (at a maximum dosage of 1 mg/kg of prednisone or equivalence a day) at the screening visit which will continue to be administered at the same dose throughout the screening period until BL/Visit 2. Steroid dose will be tapered from BL/Visit 2 onwards until week 9 (Visit 5). If the scleritis is still greater than 0.5+ on the grading scale, the investigators have the discretion to continue on the tapering course of steroid while the subjects are also being treated with ACTH gel.

The two treatment arms are as follows:

1. Mandatory 80 U twice weekly treatment with SC ACTH gel, starting at the Baseline visit (Day 0) until end of week 16.
2. Mandatory 80 U thrice weekly treatment with SC ACTH gel, starting at the Baseline visit (Day 0) until end of week 16.

Starting at week 17, treatment regimen will be determined according to clinical response to treatment as follows:

1. No evidence of active disease/disease resolved - treatment dose will be reduced to 80 U once a week with SC ACTH gel.
2. Evidence of disease improvement, but still active/partial response - ACTH treatment will continue alone at the pre-assigned treatment dose. Steroids will not be added to the treatment due to several side effects of the combination of the drugs.
3. No evidence of improvement/disease progression - treatment with ACTH gel will be discontinued and rescue therapy will be initiated as per investigator based on standard of care.

At the primary end point (week 16) and at the end of follow-up period (week 52) efficacy will be assessed by standard ophthalmic examination procedures and response to treatment, which will be graded according to established scleritis grading scale. Evaluation of response will be based on changes in scleral inflammation grade at various time points during the study, changes in pain grade scale at various time points during the study, changes in the dosage of prednisone required to maintain disease quiescence and stability and changes on ancillary testing such as FA, OCT, among others. Retreatment will be offered to study subjects who have demonstrated any level of response during the first 16 weeks and who meet any of the Retreatment Criteria listed below. Subjects receiving retreatment will receive the dose that was assigned to them at randomization. There is no placebo arm in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age ≥ 18 years;
* Able to give informed consent and attend all study visits;
* Have diagnosis of non-necrotizing scleritis determined by the Investigator to be non-infectious;
* Have active scleirits, defined as:
* Characteristic clinical presentation of active disease: painful inflammation, edema and tenderness to touch radiating to the forehead, the brow, the jaw, or the sinuses. Severity of pain associated with scleritis will be based on pain intensity, NRS scale.
* Scleral inflammation ranging from +1 to +3 as assessed by central reading center based on standardized scleritis grading scale.

and:

* are receiving no other treatment; or,
* are receiving prednisone (or equivalent dose of another corticosteroid) and/or at least 1 other systemic immunosuppressant;
* Have anterior scleritis.
* Sufficient inflammation to require systemic treatment or long-term regional treatment.
* Subjects whom the investigators feel may only need short-term topical therapy should not be enrolled.
* Best-corrected visual acuity (ETDRS method) of 20/20 to 20/400 in the study eye;
* Best- corrected visual acuity (ETDRS method) of 20/400 or better in the fellow eye
* Must have a chest radiograph within 3 months prior to enrollment with no evidence of malignancy, infection or fibrosis.
* Females of childbearing potential must have a negative urine pregnancy test at screening. In addition, sexually active females of childbearing potential must agree to use TWO of the following adequate forms of contraception while on study medication: oral, injectable, or implantable hormonal contraceptives; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner.
* Males must agree to use barrier contraception (latex condoms) when engaging in sexual activity while on study medication and for 28 days after taking the last dose of study medication.
* Prior to study screening, potential subjects must have been evaluated and screened for infectious etiologies by the investigators, possibly as part of standard clinical acre; all testing to rule out infectious causes must be performed within 3 months of screening for the ATLAS study.
* Currently active and uncontrolled scleritis, that at the determination of the investigator, requires the initiation of corticosteroid monotherapy (or equivalent), or prednisone therapy and immunomodulatory therapy or injections of corticosteroid (periocular); or scleritis in subjects for whom oral corticosteroid is contraindicated, relatively or absolutely.
* Evidence of active non-infectious scleral inflammation that at the determination of investigator requires therapy. Such evidence can be documented by clinical examination, photography, or ancillary testing (e.g. B-scan ultrasonography, fluorescein angiography, optical coherence tomography). As long as the investigator determines that the degree of inflammation can be monitored for regression or progression, the inflammation criterion can be met.
* Not planning to undergo elective ocular surgery during the first 6 months of the study.
* Subjects who have developed scleritis as ocular manifestation of an underlying systemic disease can be enrolled in the study only if the systemic therapy will not be altered throughout the study span. If at any point during the study, the ongoing systemic therapy needs to be altered (e.g. increase in the dose), the subject will have to exit the study.
* If scleritis is the initial manifestation of an underlying systemic disease, and the subjects need to be started on systemic therapy in the form of corticosteroids or immunomodulatory therapy for the underlying disease, then the subjects will not be eligible to participate in the study.
* Subjects with any or all of the following ocular complications associated with or secondary to scleritis may also be eligible for enrollment:
* Evidence of active anterior uveitis (defined as +1 cells or more in the anterior chamber or evidence of anterior vitreous inflammation on slit-lamp examination at presentation).
* Ocular hypertension, defined as intraocular pressure of ≥ 21 mmHg.
* Peripheral keratitis; defined as peripheral interstitial keratitis or thinning with either ulcerative or non-ulcerative component.10
* Subjects who have been on immunomodulatory therapy (IMT) prior to enrollment may participate in the study if they have been on a stable dose of IMT (at least 4 weeks with no change in IMT dosing or addition of new IMT agents).

Exclusion Criteria:

* Any significant ocular disease that could compromise vision in the study eye. These include, but are not limited to:

  * Diabetic retinopathy: proliferative diabetic retinopathy (PDR) or non-proliferative diabetic retinopathy (NPDR) that compromise the vision.
  * Age-related macular degeneration;
  * Myopic degeneration with active subfoveal choroidal neovascularization.
  * Advanced glaucoma status post trabeculectomy or tube/valve placement
* Any of the following treatments within 90 days prior to Day 0 or anticipated use of any of the following treatments to the study eye:

  * Intravitreal injections (including but not limited to steroids or anti-vascular endothelial growth factors);
  * Posterior subtenon's steroids.
* Intraocular surgery within 90 days prior to Day 0 in the study eye;
* Capsulotomy within 30 days prior to Day 0 in the study eye;
* Any known ocular surgery (including cataract extraction or capsulotomy) of the study eye anticipated within the first 180 days following Day 0;
* Presence of posterior scleritis as the only type of scleritis (without concurrent presence of any type of anterior scleritis;
* Intraocular pressure ≥25 mmHg in the study eye (glaucoma subjects maintained on no more than 2 topical medications with IOP <25 mmHg are allowed to participate);
* Pupillary dilation inadequate for quality stereoscopic fundus photography in the study eye;
* Media opacity that would limit clinical visualization;
* Presence of any form of ocular malignancy in the study eye, including choroidal melanoma;
* History of herpetic infection in the study eye or adnexa;
* Presence of known active or inactive toxoplasmosis in either eye;
* Presence of ocular or periocular infection in either eye;
* Participation in other investigational drug or device clinical trials within 30 days prior to Day 0, or planning to participate in other investigational drug or device clinical trials within 180 days following Day 0. This includes both ocular and non-ocular clinical trials.
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
* Prior treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples are CAMPATH, anti-CD4, anti-CD5, anti¬CD3, anti-CD19 and anti- CD20.
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline.
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline.
* Previous treatment with ACTH within 3 months of day 0 of study visit.
* Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation.

Exclusions for General Safety:

* History of severe allergic or anaphylactic reactions to proteins of porcine origin.
* Evidence of serious uncontrolled concomitant cardiovascular (including history of congestive heart failure, uncontrolled hypertension), nervous system (include myasthenia gravis), pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (includeAdrenocortical hyperfunction and primary adrenocortical insufficiency, uncontrolled diabetes mellitus, hypothyroidism), gastrointestinal disease (including history of or presence peptic ulcer disease, complicated diverticulitis, ulcerative colitis, or Crohn's disease), Scleroderma or Osteoporosis.
* Current liver disease as determined by principal investigator unless related to primary disease under investigation.
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds).
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
* Active TB requiring treatment within the previous 3 years. Subjects should be evaluated for latent and/or active TB within one month of the screening as part of the evaluation by the investigator to rule out infectious scleritis or uveitis before referring the patient to the study. If positive, subjects should be managed following local practice guidelines prior to initiating ACTH Gel. Subjects treated for TB with no recurrence in 3 years are permitted.
* Primary or secondary immunodeficiency (history of or currently active)
* Evidence of active malignant disease, malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured).
* Pregnant women or nursing (breast-feeding) mothers.
* Subjects with reproductive potential not willing to use an effective method of contraception.
* History of alcohol, drug or chemical abuse within 1 year prior to screening.
* Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation.

Laboratory Exclusion Criteria (at screening):

* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times upper limit of normal (ULN)
* Total Bilirubin> 2 times ULN
* HbA1c > 10.0 %
* White Blood Cells < 3.0 x 109/L (3000/mm3)
* Absolute Neutrophil Count < 2.0 x 109/L (2000/mm3)
* Absolute Lymphocyte Count < 0.5 x 109/L (500/mm3)
* TSH > 4U/ml or greater than normal cut-off for the lab conducting the test
* BMD (Bone Mineral Density) < -2.5 T score

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-08 (Estimated); Study Completion 2024-12-08 (Estimated)

PRIMARY OUTCOMES:
Change in grade of pain on an 11-point pain intensity numerical rating scale (NRS). | At the primary end point (week 16) and at the end of follow-up period (week 52) or at time of rescue
  The proportion of subjects demonstrating improvement (mean change from BL) by 5 points in pain, graded on an 11-point pain intensity numerical rating scale (NRS).
Change in degree of inflammation, based on the standardized scleritis grading scale. | At the primary end point (week 16) and at the end of follow-up period (week 52) or at time of rescue
  The proportion of subjects demonstrating improvement (mean change from BL) in inflammation (equal to or less than +0.5), based on the standardized scleritis grading scale.

SECONDARY OUTCOMES:
Best corrected visual acuity outcome | At week 16 (primary end point) and week 52 (end of follow-up) after therapy
  Mean change from Baseline (BL) in BCVA by ≥ 10 letters or 2 lines using the ETDRS method and at week 16 and week 52 after therapy or at time of rescue.
Vascular leakage outcome | At week 16 (primary end point) and week 52 (end of follow-up) after therapy
  Changes in degree of leakage on fluorescein angiogram (as assessed by centralized reading center) of the optic nerve and/or retinal vasculature from Baseline (BL) through week 16 and week 52.
Retinal thickness outcome | At week 16 (primary end point) and week 52 (end of follow-up) after therapy
  Changes in retinal thickness as demonstrated by spectral-domain optical coherence tomography (OCT), as assessed by the centralized reading center, for subjects with macular edema from Baseline (BL) through week 16 and week 52.
Scleral thickness outcome | At week 16 (primary end point) and week 52 (end of follow-up) after therapy
  Changes in scleral thickness as demonstrated by spectral-domain optical coherence tomography (OCT), as assessed by the centralized reading center, from Baseline (BL) through week 16 and week 52.
Dosage of systemic corticosteroids outcome | At week 16 (primary end point) and week 52 (end of follow-up) after therapy
  Changes in the dosage of systemic corticosteroids from Baseline (BL) through week 16 and week 52.
Response to therapy with/without systemic corticosteroids | At week 16 (primary end point) and week 52 (end of follow-up) after therapy
  Proportion of subjects successfully weaned off of steroids by the primary end point.
Changes in steroids dosage during study | At week 16 (primary end point) and week 52 (end of follow-up) after therapy
  Mean change in the dose of steroids from BL to primary end point and from BL to week 52.

OTHER OUTCOMES:
Incidence and severity of ocular adverse events (AEs) | At Baseline (BL) and monthly visits after screening
  The incidence and severity of ocular adverse events (AEs), as identified by eye examination (including BCVA testing), slit lamp biomicroscopy, optical coherence tomography OCT (anterior and posterior), anterior segment photography, fundus photography (FP) and fluorescein angiography (FA).
Incidence and severity of other AEs | At Baseline (BL) and monthly visits after screening
  The incidence and severity of other AEs, as identified by physical examinations, changes in vital signs, weight, clinical laboratory abnormalities, Electrocardiography (ECG) findings and subject reporting.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Chu, MD, Principal Investigator — Metropolitan Eye Research and Surgery Institute; Quan D Nguyen, MD, MSc, Principal Investigator — Stanford University; David K Scales, MD, Principal Investigator — Foresight Studies, LLC
Locations (3):
- United States (3):
  - Byers Eye Institute, Stanford University, Palo Alto, California
  - Metropolitan Eye Research and Surgery Institute, Palisades Park, New Jersey
  - Foresight Studies, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okhravi N, Odufuwa B, McCluskey P, Lightman S. Scleritis. Surv Ophthalmol. 2005 Jul-Aug;50(4):351-63. doi: 10.1016/j.survophthal.2005.04.001. PMID 15967190
- [Background] Sainz de la Maza M, Jabbur NS, Foster CS. Severity of scleritis and episcleritis. Ophthalmology. 1994 Feb;101(2):389-96. doi: 10.1016/s0161-6420(94)31325-x. PMID 8115160
- [Background] Sainz de la Maza M, Molina N, Gonzalez-Gonzalez LA, Doctor PP, Tauber J, Foster CS. Clinical characteristics of a large cohort of patients with scleritis and episcleritis. Ophthalmology. 2012 Jan;119(1):43-50. doi: 10.1016/j.ophtha.2011.07.013. Epub 2011 Oct 2. PMID 21963265
- [Background] Akpek EK, Thorne JE, Qazi FA, Do DV, Jabs DA. Evaluation of patients with scleritis for systemic disease. Ophthalmology. 2004 Mar;111(3):501-6. doi: 10.1016/j.ophtha.2003.06.006. PMID 15019326
- [Background] Keino H, Watanabe T, Taki W, Nakashima C, Okada AA. Clinical features and visual outcomes of Japanese patients with scleritis. Br J Ophthalmol. 2010 Nov;94(11):1459-63. doi: 10.1136/bjo.2009.171744. Epub 2010 Jun 24. PMID 20576778
- [Background] Erkanli L, Akova YA, Guney-Tefekli E, Tugal-Tutkun I. Clinical features, prognosis, and treatment results of patients with scleritis from 2 tertiary eye care centers in Turkey. Cornea. 2010 Jan;29(1):26-33. doi: 10.1097/ICO.0b013e3181ac9fad. PMID 19907295
- [Background] Sainz de la Maza M, Foster CS, Jabbur NS. Scleritis associated with systemic vasculitic diseases. Ophthalmology. 1995 Apr;102(4):687-92. doi: 10.1016/s0161-6420(95)30970-0. PMID 7724185
- [Background] Raiji VR, Palestine AG, Parver DL. Scleritis and systemic disease association in a community-based referral practice. Am J Ophthalmol. 2009 Dec;148(6):946-50. doi: 10.1016/j.ajo.2009.07.021. Epub 2009 Oct 17. PMID 19837380
- [Background] Watson PG, Hayreh SS. Scleritis and episcleritis. Br J Ophthalmol. 1976 Mar;60(3):163-91. doi: 10.1136/bjo.60.3.163. PMID 1268179
- [Background] Jabs DA, Mudun A, Dunn JP, Marsh MJ. Episcleritis and scleritis: clinical features and treatment results. Am J Ophthalmol. 2000 Oct;130(4):469-76. doi: 10.1016/s0002-9394(00)00710-8. PMID 11024419
- [Background] Kolomeyer AM, Ragam A, Shah K, Do BK, Shah VP, Chu DS. Cyclo-oxygenase inhibitors in the treatment of chronic non-infectious, non-necrotizing scleritis and episcleritis. Ocul Immunol Inflamm. 2012 Aug;20(4):293-9. doi: 10.3109/09273948.2012.689075. Epub 2012 May 29. PMID 22642498
- [Background] Ragam A, Kolomeyer AM, Fang C, Xu Y, Chu DS. Treatment of chronic, noninfectious, nonnecrotizing scleritis with tumor necrosis factor alpha inhibitors. Ocul Immunol Inflamm. 2014 Dec;22(6):469-77. doi: 10.3109/09273948.2013.863944. Epub 2013 Dec 19. PMID 24354512
- [Background] Jachens AW, Chu DS. Retrospective review of methotrexate therapy in the treatment of chronic, noninfectious, nonnecrotizing scleritis. Am J Ophthalmol. 2008 Mar;145(3):487-492. doi: 10.1016/j.ajo.2007.11.010. PMID 18282493
- [Background] Kolomeyer AM, Ragam A, Shah K, Jachens AW, Tu Y, Chu DS. Mycophenolate mofetil in the treatment of chronic non-infectious, non-necrotizing scleritis. Ocul Immunol Inflamm. 2012 Apr;20(2):113-8. doi: 10.3109/09273948.2012.655398. PMID 22409564
- [Background] Star RA, Rajora N, Huang J, Stock RC, Catania A, Lipton JM. Evidence of autocrine modulation of macrophage nitric oxide synthase by alpha-melanocyte-stimulating hormone. Proc Natl Acad Sci U S A. 1995 Aug 15;92(17):8016-20. doi: 10.1073/pnas.92.17.8016. PMID 7544012
- [Background] Catania A, Lonati C, Sordi A, Carlin A, Leonardi P, Gatti S. The melanocortin system in control of inflammation. ScientificWorldJournal. 2010 Sep 14;10:1840-53. doi: 10.1100/tsw.2010.173. PMID 20852827
- [Background] Baram TZ, Mitchell WG, Tournay A, Snead OC, Hanson RA, Horton EJ. High-dose corticotropin (ACTH) versus prednisone for infantile spasms: a prospective, randomized, blinded study. Pediatrics. 1996 Mar;97(3):375-9. PMID 8604274
- [Background] Fiechtner JJ, Montroy T. Treatment of moderately to severely active systemic lupus erythematosus with adrenocorticotropic hormone: a single-site, open-label trial. Lupus. 2014 Aug;23(9):905-12. doi: 10.1177/0961203314532562. Epub 2014 May 2. PMID 24795067
- [Background] Bomback AS, Canetta PA, Beck LH Jr, Ayalon R, Radhakrishnan J, Appel GB. Treatment of resistant glomerular diseases with adrenocorticotropic hormone gel: a prospective trial. Am J Nephrol. 2012;36(1):58-67. doi: 10.1159/000339287. Epub 2012 Jun 19. PMID 22722778
- [Background] Levine T. Treating refractory dermatomyositis or polymyositis with adrenocorticotropic hormone gel: a retrospective case series. Drug Des Devel Ther. 2012;6:133-9. doi: 10.2147/DDDT.S33110. Epub 2012 Jun 11. PMID 22787386
- [Background] Mittal T, Dedhia P, Roy-Chaudhury P, Abu Jawdeh BG, Mogilishetty G, Cuffy MC, Alloway RR, Woodle ES, Govil A. Complete Remission of Post-transplantation Recurrence of Focal Segmental Glomerulosclerosis With the Use of Adrenocorticotrophic Hormone Gel: Case Report. Transplant Proc. 2015 Sep;47(7):2219-22. doi: 10.1016/j.transproceed.2015.07.013. PMID 26361683
- [Background] Hladunewich MA, Cattran D, Beck LH, Odutayo A, Sethi S, Ayalon R, Leung N, Reich H, Fervenza FC. A pilot study to determine the dose and effectiveness of adrenocorticotrophic hormone (H.P. Acthar(R) Gel) in nephrotic syndrome due to idiopathic membranous nephropathy. Nephrol Dial Transplant. 2014 Aug;29(8):1570-7. doi: 10.1093/ndt/gfu069. Epub 2014 Apr 8. PMID 24714414
- [Background] Simsarian JP, Saunders C, Smith DM. Five-day regimen of intramuscular or subcutaneous self-administered adrenocorticotropic hormone gel for acute exacerbations of multiple sclerosis: a prospective, randomized, open-label pilot trial. Drug Des Devel Ther. 2011;5:381-9. doi: 10.2147/DDDT.S19331. Epub 2011 Jul 11. PMID 21792296
- [Background] Olsen NJ, Decker DA, Higgins P, Becker PM, McAloose CA, Benko AL, Kovacs WJ. Direct effects of HP Acthar Gel on human B lymphocyte activation in vitro. Arthritis Res Ther. 2015 Oct 27;17:300. doi: 10.1186/s13075-015-0823-y. PMID 26507974
- [Background] Sen HN, Sangave AA, Goldstein DA, Suhler EB, Cunningham D, Vitale S, Nussenblatt RB. A standardized grading system for scleritis. Ophthalmology. 2011 Apr;118(4):768-71. doi: 10.1016/j.ophtha.2010.08.027. Epub 2010 Nov 20. PMID 21093921
- [Background] Krebs EE, Carey TS, Weinberger M. Accuracy of the pain numeric rating scale as a screening test in primary care. J Gen Intern Med. 2007 Oct;22(10):1453-8. doi: 10.1007/s11606-007-0321-2. Epub 2007 Aug 1. PMID 17668269
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Tuft SJ, Watson PG. Progression of scleral disease. Ophthalmology. 1991 Apr;98(4):467-71. doi: 10.1016/s0161-6420(91)32269-3. PMID 2052300
- [Background] McCluskey PJ, Watson PG, Lightman S, Haybittle J, Restori M, Branley M. Posterior scleritis: clinical features, systemic associations, and outcome in a large series of patients. Ophthalmology. 1999 Dec;106(12):2380-6. doi: 10.1016/S0161-6420(99)90543-2. PMID 10599675
- [Background] Getting SJ. Targeting melanocortin receptors as potential novel therapeutics. Pharmacol Ther. 2006 Jul;111(1):1-15. doi: 10.1016/j.pharmthera.2005.06.022. Epub 2006 Feb 20. PMID 16488018
- [Background] Montero-Melendez T. ACTH: The forgotten therapy. Semin Immunol. 2015 May;27(3):216-26. doi: 10.1016/j.smim.2015.02.003. Epub 2015 Feb 26. PMID 25726511
- [Background] Brzoska T, Luger TA, Maaser C, Abels C, Bohm M. Alpha-melanocyte-stimulating hormone and related tripeptides: biochemistry, antiinflammatory and protective effects in vitro and in vivo, and future perspectives for the treatment of immune-mediated inflammatory diseases. Endocr Rev. 2008 Aug;29(5):581-602. doi: 10.1210/er.2007-0027. Epub 2008 Jul 8. PMID 18612139
- [Background] Xing Y, Parker CR, Edwards M, Rainey WE. ACTH is a potent regulator of gene expression in human adrenal cells. J Mol Endocrinol. 2010 Jul;45(1):59-68. doi: 10.1677/JME-10-0006. Epub 2010 May 11. PMID 20460446
- [Background] Manna SK, Aggarwal BB. Alpha-melanocyte-stimulating hormone inhibits the nuclear transcription factor NF-kappa B activation induced by various inflammatory agents. J Immunol. 1998 Sep 15;161(6):2873-80. PMID 9743348
- [Background] Ichiyama T, Campbell IL, Furukawa S, Catania A, Lipton JM. Autocrine alpha-melanocyte-stimulating hormone inhibits NF-kappaB activation in human glioma. J Neurosci Res. 1999 Dec 1;58(5):684-9. PMID 10561696
- [Background] Catania A, Gatti S, Colombo G, Lipton JM. Targeting melanocortin receptors as a novel strategy to control inflammation. Pharmacol Rev. 2004 Mar;56(1):1-29. doi: 10.1124/pr.56.1.1. PMID 15001661
- [Background] Lee DJ, Taylor AW. Following EAU recovery there is an associated MC5r-dependent APC induction of regulatory immunity in the spleen. Invest Ophthalmol Vis Sci. 2011 Nov 17;52(12):8862-7. doi: 10.1167/iovs.11-8153. PMID 21989727
- [Background] Lee DJ, Taylor AW. Both MC5r and A2Ar are required for protective regulatory immunity in the spleen of post-experimental autoimmune uveitis in mice. J Immunol. 2013 Oct 15;191(8):4103-11. doi: 10.4049/jimmunol.1300182. Epub 2013 Sep 16. PMID 24043903